CLINICAL TRIAL: NCT05308667
Title: Effects of Intermittent Theta Burst Stimulation in Addition to Constraint-Induced Movement Therapy in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Researcher, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulMU64
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iTBS + mCIMT group (Experimental)
  Interventions: Other: Rehabilitation (modified constraint-induced movement therapy); Other: non-invasive brain stimulation (intermittent theta-burst stimulation)
- Sham iTBS+ mCIMT group (Sham Comparator)
  Interventions: Other: Rehabilitation (modified constraint-induced movement therapy); Other: non-invasive brain stimulation (intermittent theta-burst stimulation)
- mCIMT group (Active Comparator)
  Interventions: Other: Rehabilitation (modified constraint-induced movement therapy)

INTERVENTIONS:
Other: Rehabilitation (modified constraint-induced movement therapy) — Modified constraint-induced movement therapy (mCIMT): It is an intervention used to improve functionality and mobility in the more affected upper extremity post-stroke.
Other: non-invasive brain stimulation (intermittent theta-burst stimulation) — Intermittent theta-burst stimulation (iTBS): It is a form of repetitive transcranial magnetic stimulation and it increases the facilitation of the motor cortex.
  Arms: Sham iTBS+ mCIMT group; iTBS + mCIMT group

SUMMARY:
In recent studies, it has been reported that intermittent theta-burst stimulation (iTBS) provides additional benefits when applied in adjunct to the rehabilitation in all stages of stroke (acute, subacute, or chronic). In our study, it was aimed to evaluate the effectiveness of iTBS applied in addition to modified constraint-induced movement therapy (mCIMT). By doing so, we intend to increase patient adherence to neurorehabilitation and decrease the cost of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* First time and unilateral stroke
* 1-12 months after the incident
* Getting 24 points or more in Mini Mental Status Examination
* Being able to stand for 2 minutes without any help by using the upper extremity as a support tool when necessary.
* Being a low-functioning patient according to the CIMT criteria: a) At least 10 degrees of active wrist extension starting from the angle of full flexion, b) 10 degrees of extension at the metacarpophalangeal and inter-phalangeal joints of at least 2 fingers

Exclusion Criteria:

* those who score more than 2.5 points on the Motor Activity Log-28 scale,
* who have severe pain in the upper extremity (5 and above on the Visual Analogue Scale) and spasticity (3 and above on the Modified Ashworth Scale), which may affect the treatment, and
* Those who do not have adequate communication skills.
* Patients who have visual problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper extremity | 30 minutes
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and pain.
Wolf-Motor Function Test | 45 minutes
  It is a new time-based method to evaluate upper extremity performance while providing insight into joint-specific and total limb movements

SECONDARY OUTCOMES:
Motor Evoked Potentials (MEPs) | 10 minutes
  MEPs are the electrical signals recorded from the descending motor pathways or from muscles following stimulation of motor pathways within the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersöz Hüseyinsinoğlu, Assoc. Prof., Study Director — Marmara University
Locations (1):
- Bakırköy Mazhar Osman Ruh ve Sinir Hastalıkları Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolbasi EN, Huseyinsinoglu BE, Ozdemir Z, Bayraktaroglu Z, Soysal A. Priming constraint-induced movement therapy with intermittent theta burst stimulation to enhance upper extremity recovery in patients with stroke: protocol for a randomized controlled study. Acta Neurol Belg. 2024 Jun;124(3):887-893. doi: 10.1007/s13760-024-02472-6. Epub 2024 Feb 8. PMID 38329642